CLINICAL TRIAL: NCT06817928
Title: Evaluation of the AudioKey 3 App
Brief Title: Investigating the Performance and Safety of the AudioKey 3, a Device That Provides Remote Control Options and Status Information for Compatible MED-EL Audio Processors, by Analyzing Data Logged by the App and Responses to a User Survey
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AKEY3_MED-EL_CRD_2024_03
Record Dates: First submitted 2025-01-30; First posted 2025-02-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigating the performance and safety of the AudioKey 3, a device that provides remote control options and status information for compatible MED-EL audio processors, by analyzing data logged by the app and responses to a user survey.

ELIGIBILITY:
Inclusion Criteria:

* MED-EL CI and audio processor users
* MED-EL AudioKey 3 users

Exclusion Criteria:

* Lack of compliance with any inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MED-EL CI and audio processor users MED-EL AudioKey 3 users
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
The primary objective of this clinical investigation is to confirm the performance of the AudioKey 3 app as assessed by a user survey | At time of device use
  The primary objective of this clinical investigation is to confirm the performance of the AudioKey 3 app as assessed by a user survey

SECONDARY OUTCOMES:
App user ratings obtained via user survey | At time of device use
App usage time obtained from data logging information | up to 12 months
Audio processor use obtained from data logging information | up to 12 months
• Type of implants, audio processors, auditory scenes (e.g. speech in quiet or noise) obtained from data logging information | up to 12 months
Device-related complications collected via user survey | At time of device use

CONTACTS AND LOCATIONS:
Locations (1):
- MED-EL Elektromedizinische Geräte GmbH, Innsbruck, Austria